CLINICAL TRIAL: NCT00162188
Title: Canadian Sustiva Oral Liquid Expanded Access Program: An Open-Label, Multicenter Expanded Access Study of the Liquid Formulation of Sustiva (Efavirenz, DMP266)
Brief Title: An Expanded Access Study of Oral Liquid Efavirenz in the Treatment of Children With HIV Infection: Canada
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI266-914
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

INTERVENTIONS:
Drug: Efavirenz — Oral Solution, Oral 200 - 600 mg (weight based), once daily. Until further treatment with Sustiva Oral Solution is not warranted.
  Other Names: Sustiva; BMS-561525

SUMMARY:
This study is being conducted to assess the safety and tolerability of an oral liquid solution of Sustiva for antiretroviral therapy-naive or therapy-experienced HIV-1 infected children between the ages of 3-16 who are failing or intolerant of their current antiretroviral regimen and who are unable to swallow Sustiva capsules.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-16 years of age
* Anti-retroviral naive or experienced
* Failing or intolerant to current anti-retroviral (ARV) regimen
* Limited available viable therapeutic options
* Inability to take capsules/tablets

Exclusion Criteria:

* Weighs less than 10 kg
* Failure on or concomitant use of other non-nucleoside reverse transcriptase inhibitors (NNRTIs)
* An active AIDS-defining opportunistic infection or disease
* More than two episodes of moderate to severe diarrhea or vomiting lasting more than four days within the past three months

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx